CLINICAL TRIAL: NCT07254689
Title: A Produce Prescription Program Aimed at Reducing Food Insecurity and Type 2 Diabetes Risk Among Native American Older Adults
Brief Title: The Food for Health Study
Acronym: F4H
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Maja Pedersen, Assistant Professor, University of Montana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 58394712; P20GM130418 (NIH)
Record Dates: First submitted 2025-09-24; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes; Food Insecurity; Rural Health
Keywords: produce prescription program; Native American
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Food for Health Healthy Food Prescription Intervention Arm (Experimental)
  Interventions: Behavioral: Produce Prescription Program

INTERVENTIONS:
Behavioral: Produce Prescription Program — Produce Prescription Programs (PPPs) are an upstream evidence-based intervention (EBI) to reduce food insecurity and improve health. PPPs connect healthcare services (via provider prescriptions) to vouchers for free healthy food at Food Resource Centers (FRC) to enhance access and promote healthy eating among patients. For this study the PPP will be referred to as The Food for Health (F4H) intervention and will use a clinic-to-community model to link a tribal health dept. (THD) to a local FRC through the development of new collaboration and programming. The clinic-to-community model builds local capacity for synergy across healthcare and community-based entities to address unmet health and social needs.

SUMMARY:
The project, called Food for Health (F4H), will study a new Produce Prescription Program (PPP) designed for rural Native American older adults. The study is based in the Confederated Salish and Kootenai Tribes (CSKT) of the Flathead Indian Reservation in Montana. In this community, many older adults face food insecurity and higher risk for Type 2 Diabetes (T2D). The tribal health department (THD) and local Food Resource Center (FRC) already provide important health and food support services, and this project builds on these strengths.

Produce Prescription Programs (PPPs) is a type of nutrition support intervention that connects healthcare providers with local food programs to help patients access fresh, healthy foods. For example, an individual enrolled in the study will be "prescribe" fruits and vegetables in the form of a vouchers or coupons, which can be used to buy these foods at local food centers. Research shows that this type of program can reduce food insecurity, improve diet, and support better health. PPPs also fit well with tribal community priorities by supporting food sovereignty, culture-based nutrition education, and a stronger local food system.

A key part of the study approach is using Community-Based Participatory Research (CBPR). CBPR means that community members, health providers, and researchers work together as equal partners. This way, the program is not just designed "for" the community, but "with" the community. The CSKT THD and community members have been involved in shaping this project from the start, and their priorities-like food security and food sovereignty-are at the center of the work.

The investigators will carry out the study in two phases.

Phase 1: Investigators will pilot test the acceptability of F4H in a small group of older adults (N=10) to understand the program's acceptability. The results will be used to refine and improve the program before moving to the next phase.

Phase 2: Investigators will test the feasibility and impact of the refined F4H program with a larger group of older adults (N=33). Participant food insecurity and T2D risk factors, such as blood sugar and weight, will be measured before and after the program. Investigators expect that participants will have less food insecurity and healthier measures after completing the program.

The clinic-to-community model is central to F4H. The THD will provide the prescriptions, and the FRC will be where participants redeem vouchers for fruits, vegetables, and other nutritious foods. The program will also include nutrition education that is grounded in Native culture and values. This model helps strengthen connections between healthcare and community services, creating a more supportive system for older adults.

In addition to testing the program, investigators will study how it is carried out. This is called implementation research. It means paying attention to how the program fits into the community setting, what helps it succeed, and what barriers might need to be addressed. Understanding these factors is important so that the program can continue in the future and potentially be expanded to other Native communities.

The long-term goal of F4H is to empower Native American communities to improve nutrition and reduce health disparities. By supporting older adults in gaining better access to healthy foods, the aim is to lower diabetes risk, improve quality of life, and strengthen local food systems. If the program is successful, it can serve as a model for other rural communities facing similar challenges.

DETAILED DESCRIPTION:
Study Design - Food for Health (F4H)

Type 2 diabetes (T2D) and food insecurity disproportionately affect Native American (NA) populations. These inequities are closely tied to the social determinants of health (SDOH), including limited access to affordable, nutritious foods. Food insecurity among NAs is approximately 20% higher than among non-Hispanic Whites, reflecting structural inequities rooted in the long-term impacts of colonization, forced relocation, and the disruption of traditional food systems. In response, many tribal communities are prioritizing food sovereignty, food security, and culturally relevant health interventions to address these disparities.

Produce Prescription Programs (PPPs) represent an evidence-based intervention (EBI) that directly addresses food insecurity by linking higher risk patients with access to healthy foods. Through provider-issued prescriptions, patients receive vouchers redeemable at local food outlets for fruits, vegetables, and other nutritious items. PPPs reduce barriers to healthy eating, improve diet quality, and demonstrate promise in reducing risk for chronic disease. Importantly, PPPs align well with NA community priorities to strengthen local food systems and advance culture-centered nutrition education. However, little research has examined PPP effectiveness among rural NA older adults, a critical gap given their elevated risk for T2D and underrepresentation in nutrition and implementation research.

The Food for Health (F4H) intervention aims to fill this gap. F4H is a clinic-to-community PPP designed for rural NA older adults and co-developed with the Confederated Salish and Kootenai Tribes (CSKT) of the Flathead Indian Reservation in Montana. The intervention will connect the tribal health department (THD) with a local Food Resource Center (FRC) to enhance access to fresh produce and strengthen community-based nutrition supports. A unique feature of this study is its community-based participatory research (CBPR) framework, which ensures that the intervention is designed, implemented, and evaluated in collaboration with community partners and responsive to tribal priorities such as food security and sovereignty.

The study will be conducted in two phases.

Phase 1 (Aim 1): Assess the acceptability of F4H and identify implementation determinants. Ten older adult participants (N=10) will engage in the intervention, and ten key informants (N=10) from the THD and FRC will participate in interviews. Data will provide insight into participant experiences, cultural appropriateness, and organizational readiness. Results will refine the intervention protocol and implementation plan to ensure alignment with community needs and context.

Phase 2 (Aim 2): Evaluate the feasibility, implementation strategies, and preliminary effectiveness of the refined F4H intervention in a larger sample of rural NA older adults (N=33). Key outcomes include changes in food insecurity and T2D risk factors (e.g., weight, blood glucose) measured pre- and post-intervention. Investigators hypothesize that participants will experience reduced food insecurity and improved T2D risk indicators immediately following the intervention.

The F4H model will be studied using implementation research methods, which prioritize understanding how EBIs can be integrated into real-world public health practice. This includes assessing contextual facilitators and barriers, stakeholder engagement, and sustainability potential. By embedding F4H in existing community and healthcare infrastructure, the project builds capacity for long-term impact and scalability within NA communities.

The long-term goal of this research is to empower rural NA communities to strengthen food systems, enhance access to healthy foods, and reduce the disproportionate burden of T2D among older adults. By combining evidence-based intervention strategies with a CBPR framework, this study addresses a significant gap in nutrition and implementation research and provides a foundation for larger-scale trials. If effective, F4H has the potential to serve as a scalable model for addressing food insecurity and chronic disease prevention in tribal communities nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 55 years or older
* Live on the Flathead Reservation
* Self-identify as Native American (NA)
* Food insecurity, as determined using Hunger Vital Sign™, a two question screener asked by providers.
* Pre-diabetic, based on HbA1c lab results of (5.7-6.4%) or scores 5+ on the National Diabetes Prevention Programs screener based on health and history.

Exclusion Criteria:

* Individuals with prevalent diabetes
* Individuals with end-stage renal disease
* Their health provider states they should not participate
* If a participant is unable to communicate due to severe hearing loss or speech disorder, or severe visual impairment precluding them from completing assessment.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02-15 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility Measure | Time Frame: Pre (week 0), mid (week 8), post intervention (week 17)
  A brief 5-minute Likert-style survey including items for Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM). Each scale includes five items and has demonstrated content, discriminant, and structural validity, as well as reliability and responsiveness to change.
  AIM (Acceptability): Rates the extent to which the intervention is viewed as agreeable or satisfactory (e.g., "F4H meets my approval").
  IAM (Appropriateness): Assesses the perceived fit or suitability of the intervention (e.g., "F4H seems suitable").
  FIM (Feasibility): Evaluates the extent to which the intervention can be successfully carried out (e.g., "F4H seems doable").
  Mean scores are calculated across all items and averaged together for a composite score. Higher values indicating better outcomes, with a score of 3 or higher indicating that participants view the intervention as feasible.

SECONDARY OUTCOMES:
U.S. Household Food Security Survey Module: Six-Item Short Form | Pre (week 0), mid (week 8), post intervention (week 17)
  Food security will be measured using the U.S. Household Food Security Survey Module: Six-Item Short Form (USDA, 2012). Participants respond to six questions assessing food access and affordability over the past 12 months. Affirmative responses are summed for a total score ranging from 0 to 6, with higher scores indicating greater food insecurity. Scores are categorized as high/marginal (0-1), low (2-4), or very low (5-6) food security and as binary categories, food secure (0-1) and food insecure (2-6).
  Assessments will occur via REDCap surveys. The binary outcome (secure vs. insecure), investigators will use a logistic model with pairwise comparisons.

OTHER OUTCOMES:
Glycated Hemoglobin (HbA1c) | Pre (week 0), mid (week 8), post intervention (week 17)
  Eligibility Criteria: At-Risk for Type 2 Diabetes (HbA1c or National DPP Screener)
  Eligible individuals must be classified as at risk for Type 2 Diabetes (T2D) based on one of the following criteria:
  Glycated Hemoglobin (HbA1c): A laboratory-measured HbA1c value between 5.7% and 6.4%, indicating prediabetes risk according to American Diabetes Association guidelines.
  National Diabetes Prevention Program (DPP) Screener: A score of 5 or higher on the CDC's National DPP Risk Test, based on self-reported health and lifestyle history.
  Glycated Hemoglobin (HbA1c):
  HbA1c will be measured using standardized laboratory procedures. HbA1c is reported as a percentage, scores range from normal (<5.7%), prediabetes (5.7-6.4%), to diabetes (≥6.5%). Lower scores indicate better glycemic control. Continuous HbA1c values will be analyzed using a repeated measures ANOVA to examine within-participant changes across three time points (pre, mid, post) for one treatment group.
NCI Dietary Screener Questionnaire for Fruit & Vegetable Intake | Pre (week 0), mid (week 8), post intervention (week 17)
  Self-reported fruit and vegetable (F&V) consumption will be collected using the NCI Dietary Screener Questionnaire, and will be administered via REDCap. This 10-item survey uses a 30-day reference period, converted to daily cup equivalent estimates of F&V intake
  Scores are treated as a continuous variable, with higher values indicating greater intake and, therefore, a more favorable dietary outcome. Changes across time points will be analyzed using a repeated measures ANOVA for within-subject comparisons across the three assessment periods.

IPD SHARING:
Plan to Share IPD: No
The IPD will be shared based on the data sovereignty protocol developed by the Confederated Salish and Kootenai Tribes Research Review Board.